CLINICAL TRIAL: NCT03653091
Title: Randomized, Double-Blind, Sham-Controlled, Prospective, Multi-Center Pilot Study to Evaluate the Safety and Effectiveness of Duodenal Mucosal Resurfacing Using the Revita™ System in the Treatment of Type 2 Diabetes
Brief Title: Safety & Effectiveness of Duodenal Mucosal Resurfacing (DMR) Using the Revita™ System in Treatment of Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fractyl Health Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-40000
Record Dates: First submitted 2018-08-24; First posted 2018-08-31 (Actual); Results first posted 2022-07-26 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; Diabetes Mellitus; Noninsulin-Dependent Diabetes Mellitus; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases; Revita System; Anti-diabetic medications; Duodenal Mucosal Resurfacing
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Duodenal Mucosal Resurfacing (DMR) (Active Comparator): Duodenal Mucosal Resurfacing (DMR) treatment will include hydrothermal ablation of the duodenal mucosa in an upper endoscopic procedure in patients with type 2 diabetes.
  Interventions: Device: Duodenal Mucosal Resurfacing (DMR)
- Duodenal Mucosal Resurfacing Sham (Sham) (Sham Comparator): Duodenal Mucosal Resurfacing Sham (Sham) treatment will include an upper endoscopic procedure similar to DMR treatment without hydrothermal ablation of the duodenal mucosa in patients with type 2 diabetes.
  Interventions: Device: Duodenal Mucosal Resurfacing Sham (Sham)

INTERVENTIONS:
Device: Duodenal Mucosal Resurfacing (DMR) — The Fractyl DMR procedure utilizes the Revita™ Catheter to perform hydrothermal ablation of the duodenum. The catheter is delivered trans-orally over a guide-wire to first inject saline to lift the sub-mucosal space, followed by an ablation of the duodenal mucosa. Subjects who receive the DRM treatment are followed for 48 weeks while Sham subjects who cross over and undergo the DMR procedure at 24 weeks are followed for further 24 weeks post treatment. Sham subjects who choose not to cross over are discontinued from the study.
  Arms: Duodenal Mucosal Resurfacing (DMR)
Device: Duodenal Mucosal Resurfacing Sham (Sham) — The Sham procedure consists of placing the Revita™ Catheter as described above into the duodenum for a minimum of 30 minutes and then removing it from the patient.
  Arms: Duodenal Mucosal Resurfacing Sham (Sham)

SUMMARY:
The Revita™ System is being investigated to assess the ability to improve glycemic control in conjunction with diet and exercise in patients with Type 2 diabetes who are inadequately controlled with oral anti-diabetic medications. The purpose of this study is to demonstrate the safety and effectiveness of the Fractyl DMR Procedure using the Revita™ System compared to a sham procedure. At 24 weeks, subjects randomized to the DMR procedure be continued to be followed per protocol till 48 Weeks and the Sham treatment arm will be offered to cross over to receive the DMR treatment and will be followed per protocol for 24 weeks post treatment.

DETAILED DESCRIPTION:
The study is a randomized, double-blind sham-controlled prospective multi-center clinical investigation of subjects with T2D sub-optimally controlled on two oral anti-diabetic medications, one of which must be metformin, comparing the Fractyl DMR procedure using the Revita™ System to a sham procedure. All subjects will participate in a 4 week oral anti-diabetic medication run-in period before the procedure to confirm inadequate blood glucose control in conjunction with medication compliance and nutritional counseling. Subjects who meet all criteria after screening are randomized 2:1 (DMR to sham), with double blinding (subject and endocrinologist/Sponsor). The endoscopist is not blinded.

ELIGIBILITY:
Inclusion Criteria:

1. Men and non-pregnant women 28-65 years of age
2. Diagnosed with T2D for at least 3 years
3. A1C of 7.5 - 9.5% (59-80 mmol/mol)
4. BMI ≥ 28 and ≤ 40 kg/m2
5. On two to three oral OADs (metformin plus one to two additional OADs) with two (see note below) at least at half maximum labeled dose (or highest tolerated) with no changes in medication in the 12 weeks prior to the Screening Visit (Visit 1) (Refer to ADA Standard of Medical Care in Diabetes 2018, Table 8.3 for the maximum approved daily dose of non-insulin glucose lowering agents) (43). Note: For subjects on sulfonylurea (SU) glucose-lowering drugs for diabetes, the only SUs permitted in the study will be glipizide or glimepiride, and their doses below half maximum labeled dosing will not be an exclusion for study entry. Patients unwilling to reduce the dose of SU at the time of the DMR procedure as described by protocol will be excluded.
6. Agree to use an additional glucose-lowering treatment (eg, liraglutide, other OAD with the exception of glyburide) if recommended by the study investigator in case of persistent hyperglycemia.
7. Agree not to donate blood during their participation in the study
8. Able to comply with study requirements and understand and sign the Informed Consent Form
9. Women of childbearing potential (WOCBP) must be using two acceptable methods of contraception throughout the study
10. Women must not be breastfeeding

Exclusion Criteria:

1. Diagnosed with Type 1 Diabetes (T1D)
2. History of diabetic ketoacidosis or hyperosmolar nonketotic coma
3. Probable insulin production failure, defined as fasting C Peptide serum <1 ng/mL (333pmol/l)
4. Previous use of any types of insulin for >1 month (at any time, except for treatment of gestational diabetes)
5. Current use of injectable medications for diabetes (insulin, GLP-1RA)
6. Current use of glyburide, a sulfonylurea (SU) glucose-lowering drug for diabetes
7. Hypoglycemia unawareness or a history of severe hypoglycemia (more than 1 severe hypoglycemic event, as defined by need for third-party-assistance, in the last year)
8. Known autoimmune disease, including but not limited to celiac disease, or pre-existing symptoms of systemic lupus erythematosus, scleroderma or other autoimmune connective tissue disorder
9. Previous GI surgery that could limit treatment of the duodenum such as Bilroth 2, Roux-en-Y gastric bypass, or other similar procedures or conditions
10. History of chronic or acute pancreatitis
11. History of diabetic gastroparesis
12. Known active hepatitis or active liver disease
13. Acute gastrointestinal illness in the previous 7 days
14. Known history irritable bowel syndrome, radiation enteritis or other inflammatory bowel disease, such as Crohn's disease
15. Known history of a structural or functional disorder of the esophagus that may impede passage of the device through the gastrointestinal tract or increase risk of esophageal damage during an endoscopic procedure, including Barrett's esophagus, esophagitis, dysphagia, achalasia, stricture/stenosis, esophageal varices, esophageal diverticula, esophageal perforation, or any other disorder of the esophagus
16. Known history of a structural or functional disorder of the esophagus, including any swallowing disorder, esophageal chest pain disorders, or drug refractory esophageal reflux symptoms
17. Known history of a structural or functional disorder of the stomach including gastroparesis, gastric ulcer, chronic gastritis, gastric varices, hiatal hernia (> 2 cm), cancer or any other disorder of the stomach
18. Known history of chronic symptoms suggestive of a structural or functional disorder of the stomach, including any symptoms of chronic upper abdominal pain, chronic nausea, chronic vomiting, chronic dyspepsia or symptoms suggestive of gastroparesis, including post-prandial fullness or pain, post-prandial nausea or vomiting or early satiety
19. Known history of duodenal ulcer, intestinal diverticula (diverticulitis), intestinal varices, intestinal stricture/stenosis, small bowel obstruction, or any other obstructive disorder of the GI tract
20. Currently have ongoing symptoms suggestive of intermittent small bowel obstruction, such as recurrent bouts of post-prandial abdominal pain, nausea or vomiting
21. Active H. pylori infection (Subjects with active H. pylori may continue with the screening process if they are treated with an appropriate antibiotic regimen)
22. History of coagulopathy, upper gastrointestinal bleeding conditions such as ulcers, gastric varices, strictures, congenital or acquired intestinal telangiectasia
23. Current use of anticoagulation therapy (such as warfarin) which cannot be discontinued for 7 days before and 14 days after the procedure
24. Current use of P2Y12 inhibitors (clopidogrel, pasugrel, ticagrelor) which cannot be discontinued for 14 days before and 14 days after the procedure.
25. Unable to discontinue non-steroidal anti-inflammatory drugs (NSAIDs) during treatment through 4 weeks following the procedure. Use of low dose aspirin is allowed.
26. Current use of serotonergic medications (SSRI)
27. Use of systemic glucocorticoids (excluding topical or ophthalmic application or inhaled forms) for more than 10 consecutive days within 90 days prior to the Screening Visit
28. Use of drugs known to affect GI motility (e.g. Metoclopramide)
29. Receiving weight loss medications such as Meridia, Xenical, or over the counter weight loss medications
30. Untreated/inadequately treated hypothyroidism, defined as an elevated Thyroid-Stimulating Hormone (TSH) level at Screening; if on thyroid hormone replacement therapy, must be on stable dose for at least 6 weeks prior to Screening
31. Persistent Anemia, defined as Hemoglobin <10 g/dL
32. Subjects who have donated blood or received a transfusion in the prior 3 months
33. Subjects with conditions that alter red blood cell turnover
34. Subjects with prosthetic joints
35. Significant cardiovascular disease including known history of valvular disease, or myocardial infarction, heart failure, transient ischemic attack or stroke within the last 6 months
36. Moderate or severe chronic kidney disease (CKD), with estimated glomerular filtration rate (eGFR) <45 ml/min/1.73m2 (estimated by MDRD)
37. Known immunocompromised status, including but not limited to individuals who have undergone organ transplantation, chemotherapy or radiotherapy within the past 12 months, who have clinically-significant leukopenia, who are positive for the human immunodeficiency virus (HIV) or whose immune status makes the subject a poor candidate for clinical trial participation in the opinion of the Investigator
38. Active systemic infection
39. Active malignancy within the last 5 years (with the exception of treated basal cell or treated squamous cell carcinoma)
40. Subjects with a personal or family history of medullary thyroid carcinoma
41. Subjects with Multiple Endocrine Neoplasia syndrome type 2
42. Not a candidate for surgery or general anesthesia
43. Active illicit substance abuse or alcoholism
44. Current smoker
45. Participating in another ongoing clinical trial of an investigational drug or device
46. Any other mental or physical condition which, in the opinion of the Investigator, makes the subject a poor candidate for clinical trial participation
47. Unwilling or unable to perform SMBG, complete the patient diary, or comply with study visits and other study procedures as required per protocol

Additional exclusion criteria to be confirmed during the screening process:

1. A1c post Run-In Phase < 7.5% (59 mmol/mol) or > 9.5% (86 mmol/mol)
2. Any severe hypoglycemic event, defined as hypoglycemia requiring third-party assistance; or any clinically significant hypoglycemic event, defined as self-monitored or laboratory plasma glucose level < 54 mg/dL (3.0 mmol/L); or ≥ 2 glucose alert values ≤70 mg/dL (3.9 mmol/L), unless a clear correctable precipitating factor can be identified, since the screening visit (Visit 1)
3. Uncontrolled hyperglycemia with a glucose level >270 mg/dl (>15 mmol/L) after an overnight fast or >360 mg/dl (>20 mmol/l) in a randomly performed measurement during Medication Run-In Period and confirmed by a second measurement (not on the same day)
4. Mean of 3 separate blood pressure measurements >180 mmHg (systolic) or >100 mmHg (diastolic)
5. WOCBP with a positive urine pregnancy test at Baseline Visit
6. Active and uncontrolled GERD defined as grade III esophagitis or greater
7. Abnormalities of the GI tract preventing endoscopic access to the duodenum
8. Anatomic abnormalities in the duodenum that would preclude the completion of the DMR procedure, including tortuous anatomy
9. Malignancy newly diagnosed by endoscopy
10. Upper gastrointestinal conditions such as ulcers, polyps, varices, strictures, congenital or acquired intestinal telangiectasia

Ages: 28 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-09-28 (Actual); Primary Completion 2020-08-10 (Actual); Study Completion 2020-08-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Florida Hospital / TRANSLATIONAL RESEARCH INSTITUTE FOR METABOLISM AND DIABETES (TRI), Orlando, Florida
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - University of Pennsylvania - Penn Metabolic Medicine, Philadelphia, Pennsylvania
  - UTHealth, Houston, Texas
  - Texas Diabetes Institute, San Antonio, Texas

REFERENCES:
- [Derived] Busch CBE, Meiring S, van Baar ACG, Gastaldelli A, DeFronzo R, Mingrone G, Hagen M, White K, Rajagopalan H, Nieuwdorp M, Bergman JJGHM. Insulin sensitivity and beta cell function after duodenal mucosal resurfacing: an open-label, mechanistic, pilot study. Gastrointest Endosc. 2024 Sep;100(3):473-480.e1. doi: 10.1016/j.gie.2024.01.031. Epub 2024 Jan 25. PMID 38280531

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All eligible subjects participated in a 4-week oral antidiabetic drug (OAD) run-in period before randomization to the index procedure to assess stability of blood glucose control in conjunction with medication compliance and lifestyle (diet, exercise) counseling. All subjects were managed according to the current diabetes standard of care.
Groups:
- Duodenal Mucosal Resurfacing Procedure (DMR): Duodenal Mucosal Resurfacing (DMR) treatment will include hydrothermal ablation of the duodenal mucosa in an upper endoscopic procedure in patients with type 2 diabetes.
  The Fractyl DMR procedure utilizes the Revita™ Catheter to perform hydrothermal ablation of the duodenum. The catheter is delivered trans-orally over a guide-wire to first inject saline to lift the sub-mucosal space, followed by an ablation of the duodenal mucosa. Subjects who receive the DRM treatment are followed for 48 weeks.
- Sham Procedure (Sham): Sham treatment (Sham) will include an upper endoscopic procedure similar to DMR treatment without hydrothermal ablation of the duodenal mucosa in patients with type 2 diabetes.
  The Sham procedure consists of placing the Revita™ Catheter as described above into the duodenum for a minimum of 30 minutes and then removing it from the patient.
  Sham subjects who cross over and undergo the DMR procedure at 24 weeks are followed for further 24 weeks post treatment. Sham subjects who choose not to cross over are discontinued from the study.
Period: First 24 Weeks
Arm/Group | Duodenal Mucosal Resurfacing Procedure (DMR) | Sham Procedure (Sham)
Started | 6 | 3
Intent-to-Treat | 6 | 3
As-Treated (One participant randomized to the DMR arm received Sham, had the option to crossover, and was included in the Sham arm.) | 5 | 4
Safety | 5 | 4
Completed | 6 | 3
Not Completed | 0 | 0
Period: Second 24 Weeks
Arm/Group | Duodenal Mucosal Resurfacing Procedure (DMR) | Sham Procedure (Sham)
Started (The As-Treated population is being used) | 5 | 4
Crossed Over to DMR at Week 24 | 0 | 3
Completed | 5 | 3
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Duodenal Mucosal Resurfacing Procedure (DMR): Duodenal Mucosal Resurfacing (DMR) treatment will include hydrothermal ablation of the duodenal mucosa in an upper endoscopic procedure in patients with type 2 diabetes.
  The Fractyl DMR procedure utilizes the Revita™ Catheter to perform hydrothermal ablation of the duodenum. The catheter is delivered trans-orally over a guide-wire to first inject saline to lift the sub-mucosal space, followed by an ablation of the duodenal mucosa. Subjects who receive the DRM treatment are followed for 48 weeks while Sham subjects who cross over and undergo the DMR procedure at 24 weeks are followed for further 24 weeks post treatment. Sham subjects who choose not to cross over are discontinued from the study.
- Sham Procedure (Sham): Sham treatment (Sham) will include an upper endoscopic procedure similar to DMR treatment without hydrothermal ablation of the duodenal mucosa in patients with type 2 diabetes.
  The Sham procedure consists of placing the Revita™ Catheter as described above into the duodenum for a minimum of 30 minutes and then removing it from the patient.
- Total: Total of all reporting groups
Arm/Group | Duodenal Mucosal Resurfacing Procedure (DMR) | Sham Procedure (Sham) | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 4 | 9
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Standard Deviation); unit: years] | 57.0 (3.83) | 53.5 (4.20) | 56.0 (3.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 4 | 4 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 5 | 3 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 4 | 2 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 4 | 9
Height (cm) [Mean (Standard Deviation); unit: cm] | 171.44 (9.871) | 176.03 (5.954) | 173.48 (8.237)
Weight (kg) [Mean (Standard Deviation); unit: kg] | 92.24 (7.513) | 94.4 (7.366) | 93.2 (7.062)
Body mass index (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 31.50 (2.630) | 30.28 (1.841) | 30.96 (2.268)
HbA1c (%) [Mean (Standard Deviation); unit: mmol/mol] | 8.3 (.738) | 8.73 (.512) | 8.49 (.649)
Duration of T2D Diagnosis (days) [Mean (Standard Deviation); unit: Days] | 4222.6 (1442) | 4933 (1703.53) | 4538.3 (1506.03)

OUTCOME MEASURES:

1. Primary Outcome: Change in Hemoglobin A1c (HbA1c)
Description: Change in HbA1c from baseline in DMR vs Sham groups
Time Frame: 24 weeks post procedure
Population: The AT population is a subset of ITT subjects who received at least 1 ablation or underwent the randomized sham procedure.
Measure: Mean (Standard Deviation); unit: mmol/mol
Arm/Group | Duodenal Mucosal Resurfacing (DMR) | Duodenal Mucosal Resurfacing Sham (Sham)
Number analyzed (Participants) | 5 | 4
mmol/mol | -0.33 (.252) | -0.70 (.469)

ADVERSE EVENTS:
Time Frame: Adverse events were followed for up to a maximum of 56 weeks.
Description: Deaths and/or Adverse Events are reported using the Safety Population.
Groups:
- Sham Crossover: Subjects that were in sham arm until 24 weeks and then crossover to receive DMR treatment at 24 weeks and followed up for additional 24 weeks. AEs captured from time of DMR procedure through follow up to end of study.
Arm/Group | Duodenal Mucosal Resurfacing Procedure (DMR) | Sham Procedure (Sham) | Sham Crossover
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 4/5 | 4/4 | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Duodenal Mucosal Resurfacing Procedure (DMR) (N=5) | Sham Procedure (Sham) (N=4) | Sham Crossover (N=3)
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 2
Abdominal Distension (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Respiratory Symptom (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Nodule (General disorders) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0
Mental Status Changes (Psychiatric disorders) | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Ear Pain (Ear and labyrinth disorders) | 0 | 1 | 0
Blood Glucose Increased (Investigations) | 0 | 1 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Limitations of this pilot study include the small sample size and missing data due to COVID-19.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-07-09): https://cdn.clinicaltrials.gov/large-docs/91/NCT03653091/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-19): https://cdn.clinicaltrials.gov/large-docs/91/NCT03653091/SAP_001.pdf